CLINICAL TRIAL: NCT02661711
Title: Prospective Non-randomised Exploratory Study to Assess the Safety and Efficacy of Aflibercept (Eylea) in Cystoid Macular Oedema (CMO) Associated With Retinitis Pigmentosa (RP)
Brief Title: Aflibercept for Macular Oedema With Underlying Retinitis Pigmentosa (AMOUR) Study
Acronym: AMOUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MICM1014; 2015-003723-65 (EudraCT Number)
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Macular Oedema; Retinitis Pigmentosa
Keywords: Macular Oedema Retinitis Pigmentosa
MeSH Terms: conditions — Macular Edema; Retinitis Pigmentosa | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept (Eylea) (Experimental): All patients recruited to the study will receive 3 loading intravitreal injections of Aflibercept (Eylea) at monthly intervals followed by a treat and extend protocol up to 12 months. Extension from monthly to 6, 8, 10 and 12 week follow-up will occur when there is evidence of OCT stability in the view of the investigator i.e. there is no further reduction in macular fluid compared to the previous visit. All patients will receive 5 injections before considering them non-responders.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — 2mg of 40mg/ml of Eylea Solution administered via intravitreal injection every four weeks for three months (loading dose), followed by a treat and extend protocol up to 12 months. Extension from monthly to 6, 8, 10 and 12 week follow up will occur where there is no reduction in macula oedema compared with the previous visit.
  Number of cycles; minimum of 5 injections and maximum of 13 injections per study eye.
  Other Names: Eylea

SUMMARY:
The purpose of this study is to assess the safety and efficacy of intravitreal injections of Aflibercept (Eylea) in treating Cystoid Macula Oedema (CMO) in patients with underlying Retinitis Pigmentosa (RP).

DETAILED DESCRIPTION:
This is a 17 month phase II therapeutic exploratory trial in Cystoid Macular Oedema (CMO) with underlying Retinitis Pigmentosa (RP). The study design is a prospective, open-label, interventional non-randomised trial. All patients enrolled in the study will receive intravitreal injections of Aflibercept (Eylea).

There will be a 9 month recruitment window and patient participation will be for 12 months; 30 patients aged 16 years or older presenting in the Medical Retina and Genetics clinics at Moorfields Eye Hospital with Cystoid Macula Oedema (CMO) with underlying Retinitis Pigmentosa (RP) will be approached by the study team to discuss participation in the AMOUR study and be given a patient information leaflet. If patients decide to participate in the study they will be invited to the NIHR Moorfields Clinical Research Facility for a baseline screening where written informed consent will be given by the patient and various assessments will be performed to confirm eligibility.

Patients enrolled in the study will receive intravitreal injections of 2mg of 40mg/ml of Aflibercept (Eylea) solution in the study eye. In the first three months, patients will receive a loading dose of Aflibercept (Eylea) with one injection every four weeks. After the first three months, treatment frequency will follow a treat and extend protocol for up to 12 months from date of study enrolment. Extension from 4 weekly to 6,8,10 and 12 week follow up will occur when there is no further reduction in macula fluid compared to the previous visit. Patients will receive a minimum of 5 injections before being deemed as non-responders to treatment.

Imaging and assessments such as optical coherence tomography imaging, microperimetry and visual acuity will be used to assess response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* CMO in association with RP
* > 16 years of age
* Unilateral or Bilateral CMO (the worse eye only will be treated - defined as the eye with a greater central macular thickness (CMT) on OCT)
* No previous oral treatment for CMO for last 3 months
* No previous peribulbar or intravitreal treatment for CMO in the study eye for last 3 months
* No previous topical treatment for CMO in the study eye for last 1 month
* Central visual impairment that in the view of the Principal Investigator is due to CMO
* BCVA better than 3/60

Exclusion Criteria:

* Insufficient patient cooperation or media clarity to allow adequate fundus imaging.
* Evidence of visually significant vitreo-retinal traction or epiretinal membrane on OCT that in the Principal Investigator's opinion is highly likely to significantly limit the efficacy of intravitreal therapy.
* History of cataract surgery within prior 3 months or cataract surgery anticipated within 6 months of starting the study.
* Any anti-VEGF treatment to study eye within 3 months.
* History of YAG capsulotomy performed within 3 months.
* Uncontrolled Intraocular pressure (IOP) > = 24 mmHg for ocular hypertension (on topical IOP lowering medications)
* Advanced glaucoma (in the opinion of a glaucoma specialist).
* Patients with active or suspected ocular or periocular infections
* Patients with active severe intraocular inflammation.
* Patients with a new, untreated retinal tear or detachment
* Patients with a stage 3 or 4 macular hole
* Thromboembolic event (MI/CVA/Unstable Angina) within 6 months.
* Pregnancy or family planned within 15 months
* Females who are breast feeding
* Known allergy or hypersensitivity to anti-VEGF products

Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 12 weeks after treatment discontinuation. The MHRA advise double contraception.

Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for trial treatment.

Note: Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Michaelides, Professor, Principal Investigator — Moorfields Eye Hospital, Institute of Ophthalmology
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be disclosed publically, all the data will be anonymised and analysed in accordance with the Data Protection Act

REFERENCES:
- [Derived] Strong SA, Peto T, Bunce C, Xing W, Georgiou M, Esposti SD, Kalitzeos A, Webster A, Michaelides M. Prospective exploratory study to assess the safety and efficacy of aflibercept in cystoid macular oedema associated with retinitis pigmentosa. Br J Ophthalmol. 2020 Sep;104(9):1203-1208. doi: 10.1136/bjophthalmol-2019-315152. Epub 2020 Feb 10. PMID 32041720

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravitreal Aflibercept for RP-CMO: 30 patients recruited for this study, all of which receive the active drug, aflibercept
Period: Overall Study
Arm/Group | Intravitreal Aflibercept for RP-CMO
Started | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Central Macular Thickness (CMT) on Spectral Domain OCT (SDOCT) at 12 Months
Description: Mean Central Macular Thickness (CMT) on Spectral Domain OCT (SDOCT) at 12 months
Time Frame: at 12 months
Measure: Mean (Standard Deviation); unit: Microns
Units Other Than Participants: eyes
Groups:
- Intravitreal Aflibercept for RP-CMO: Intravitreal aflibercept for RP-CMO
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
Microns | 413.4 (98.2)

2. Secondary Outcome: The Mean Change in Central Macular Thickness on Spectral Domain Optical Coherence Tomography (SD-OCT) From Baseline to 6 Months and Baseline to 12 Months
Time Frame: baseline to 6 months and baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: Microns
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
Microns
  Mean change in CMT from baseline to 6 months | -46.2 [-87.6 to -4.9]
  Mean change in CMT from baseline to 12 months | -47.6 [-80.5 to -14.6]

3. Secondary Outcome: The Mean Best Corrected Visual Acuity (BCVA) Using the ETDRS Visual Acuity Chart at 6 and 12 Months
Description: Mean Best Corrected Visual Acuity (BCVA) using the ETDRS visual acuity chart at 6 and 12 months.
  BCVA is the best possible vision an eye can see with corrective lenses, measured using the ETDRS visual acuity chart. The ETDRS score is calculated as the total number of letters correctly read at 4m from the chart plus 30 (if 20 or more letters can be read at 4m).
Time Frame: baseline to 6 months and baseline to 12 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
ETDRS letters
  Mean BCVA at 6 months | 66.9 (10.6)
  Mean BCVA at 12 months | 68.0 (11.1)

4. Secondary Outcome: The Mean Change in ETDRS BCVA at 6 Months and at 12 Months
Description: Mean ETDRS BCVA change at 6 months and at 12 months. BCVA is the best possible vision an eye can see with corrective lenses, measured using the ETDRS visual acuity chart. The ETDRS score is calculated as the total number of letters correctly read at 4m from the chart plus 30 (if 20 or more letters can be read at 4m).
Time Frame: at 6 months and at 12 months
Measure: Mean (Standard Deviation); unit: ETDRS letters
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
ETDRS letters
  Mean change in BCVA from baseline to 6 months | 3.1 (6.6)
  Mean change in BCVA from baseline to 12 months | 4.3 (6.9)

5. Secondary Outcome: The Mean Macular Volume on SDOCT at 6 and 12 Months
Time Frame: baseline to 6 months and baseline to 12 months
Measure: Mean (Standard Deviation); unit: millimeters cubed
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
millimeters cubed
  Mean macular volume at 6 months | 7.9 (0.6)
  Mean macular volume at 12 months | 8.0 (0.7)

6. Secondary Outcome: The Mean Change in Macular Volume on SDOCT From Baseline to 6 Months and Baseline to 12 Months
Time Frame: baseline to 6 months and baseline to 12 months
Measure: Mean (Standard Deviation); unit: millimeters cubed
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
millimeters cubed
  Mean change mac volume from baseline to 6 months | -0.3 (0.8)
  Mean change mac volume from baseline to 12 months | -0.3 (0.7)

7. Secondary Outcome: Report All Adverse Events and Serious Adverse Events
Time Frame: From date of first injection for first patient to the end of the study (17 months)
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 30
Number analyzed (eyes) | 30
participants
  Non-serious adverse events in whole study | 26
  Serious adverse events in whole study | 1

8. Secondary Outcome: The Mean Retinal Sensitivity Using Microperimetry at 6 and 12 Months
Time Frame: At 6 months and at 12 months
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
decibels
  Mean retinal sensitivity at 6 months | 4.92 (3.49)
  Mean retinal sensitivity at 12 months | 4.93 (3.49)

9. Secondary Outcome: The Mean Change in Retinal Sensitivity Using Microperimetry From Baseline to 6 Months and Baseline to 12 Months
Time Frame: From baseline to 6 months and baseline to 12 months
Measure: Mean (Standard Deviation); unit: decibels
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
decibels
  Mean change ret sens from baseline to 6 months | -1.23 (2.24)
  Mean change ret sens from baseline to 12 months | -1.09 (2.10)

10. Secondary Outcome: The Mean Number of Intravitreal Injections Administered
Time Frame: 17 months (from first patient first visit to last patient last visit)
Measure: Median (Inter-Quartile Range); unit: injections
Units Other Than Participants: eyes
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
Number analyzed (eyes) | 29
injections | 7 [6 to 9]

11. Secondary Outcome: The Mean Central Macular Thickness (CMT) on Spectral Domain OCT (SDOCT) at 6 Months
Description: The Mean Central Macular Thickness (CMT) on Spectral Domain OCT (SDOCT) at 6 Months
Time Frame: at 6 months
Population: 29
Measure: Mean (Standard Deviation); unit: micron
Groups:
- Intravitreal Aflibercept for RP-CMO: Arm received Intravitreal Aflibercept for RP-CMO
Arm/Group | Intravitreal Aflibercept for RP-CMO
Number analyzed (Participants) | 29
micron | 414.8 (96.4)

ADVERSE EVENTS:
Time Frame: Up to 17 months for the study duration.
Description: Systematic collection at every patient visit
Groups:
- Aflibercept for RP-CMO: This arm received Aflibercept for RP-CMO
Arm/Group | Aflibercept for RP-CMO
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept for RP-CMO (N=30)
Sub-acute reduction of vision (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept for RP-CMO (N=30)
Ocular adverse events (Eye disorders) | 18 (39)
Systemic adverse event (General disorders) | 17 (35) — Including anything reported by the patient at any time throughout the duration of the study, for example: bad back, feeling low, viral illness, bitten by mosquito, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-11-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT02661711/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT02661711/SAP_001.pdf
  • Informed Consent Form (2016-03-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02661711/ICF_002.pdf